CLINICAL TRIAL: NCT07306910
Title: Effect of Opioid-Free Anesthesia (OFA) on Postoperative Pain and Perioperative Nausea and Vomiting in Elective Laparoscopic Cholecystectomy.
Brief Title: Effect of Opioid-Free Anesthesia (OFA) on Postoperative Pain and Perioperative Nausea and Vomiting in Elective Laparoscopic .
Acronym: OFA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Galal Eldeen Hasan Hasan Hussein, resident at the anesthesia , icu and pain management department, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 211198; 211198 (Registry Identifier: galal eldeen hasan hasan)
Record Dates: First submitted 2025-10-17; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Opioid-Free Anesthesia; Elective Laparoscopic Cholecystectomy
Keywords: opa
MeSH Terms: interventions — Lidocaine; Dexmedetomidine; Magnesium

STUDY DESIGN:
Intervention Model Description: Type of the study: Prospective, triple-blind, parallel-group, superiority block randomized controlled trial. Study Setting and design features.
  • Allocation: Computer-generated 1:1 block randomization with allocation concealment (block size = 6), stratified by ASA status (I vs II/III).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Blinding: Participants, anesthetist/ clinicians obserevers and data analysts will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OpioidSparingGroup OS) (Active Comparator)
  Interventions: Other: opoid free anesthesia
- ControlGroup (CG) (Active Comparator)
  Interventions: Other: opoid free anesthesia

INTERVENTIONS:
Other: opoid free anesthesia — Maintenance Dexmedetomidine 0.2-0.5 µg/kg/h + Lidocaine 1.5 mg/kg/h + Magnesium 10 mg/kg/h; Sevoflurane as required; Atracurium 0.1 mg/kg IV PRN
  Other Names: Lidocaine; Dexmedetomidine; Magnesium

SUMMARY:
1. To evaluate the eﬃcacy of a standardized multimodal Opioid Sparing (OS) protocol versus conventional opioid-based analgesia in reducing acute postoperative
2. To quantify opioid consumption reduction achievable through OS strategies
3. To assess the impact of OS on hemodynamic parameters during critical surgical phases
4. To compare recovery metrics (PONV, bowel function, ambulation)
5. To evaluate the safety proﬁle of OS anesthesia

DETAILED DESCRIPTION:
The ongoing opioid crisis represents a signiﬁcant public health challenge, with surgical prescriptions being a major contributor to chronic opioid use and misuse. Recent epidemiological data indicate that 4-6% of opioid- naïve patients develop persistent opioid use postoperatively, with laparoscopic cholecystectomy patients being particularly vulnerable due to moderate postoperative pain . Despite being a minimally invasive procedure, laparoscopic cholecystectomy consistently ranks among the most common general surgical procedures worldwide, with over 1 million performed annually in the United States alone. This frequency ampliﬁes the population-level impact of postoperative prescribing patterns . Previous studies have demonstrated the eﬃcacy of individual components-dexmedetomidine for hemodynamic stabilization, lidocaine infusions for visceral analgesia, and regional techniques like erector spinae plane (ESP) blocks-but their synergistic effects remain underexplored . A recent scoping review highlighted that while opioid-sparing (OS) effects are frequently reported, evidence for clinically meaningful outcomes (e.g., reduced ventilation time, accelerated functional recovery) remains limited . The pathophysiology of post-cholecystectomy pain involves both somatic (abdominal wall) and visceral (diaphragmatic irritation, biliary spasm) components, necessitating a multimodal approach. Opioids inadequately address inﬂammatory mediators while introducing risks of respiratory depression, postoperative nausea and vomiting (PONV), ileus, and hemodynamic instability. Emerging evidence suggests that α-2 agonists (e.g., dexmedetomidine) and NMDA ant

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 60 years scheduled for elective laparoscopic cholecystectomy. Elective must be included in title.
* ASA (American Society of Anesthesiologists) physical status I or II.
* Body Mass Index (BMI) < 35 kg/m².

Exclusion Criteria:

* Chronic opioid use (>30 MME/day for >3 months).
* Contraindications to study medications (e.g., severe hepatic impairment; allergy/contraindication to lidocaine, dexmedetomidine, ketamine, fentanyl, or NSAIDs).
* Renal dysfunction (eGFR <60 mL/min/1.73 m²).
* Significant cardiac conduction abnormalities.
* Pregnancy or lactation.
* Emergency surgery or conversion to open cholecystectomy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity at rest postoperatively (Visual Analog Scale, VAS, 0-10) | 48 hours post operative
  Pain intensity at rest will be measured using the Visual Analog Scale (VAS), which ranges from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate worse pain.

SECONDARY OUTCOMES:
Cumulative opioid use (MME) | 48 hours post operative
  Cumulative opioid consumption will be measured in morphine milligram equivalents (MME) administered to each patient.
Time to extubating | 24 hours post operative
  Time to extubating; time to Aldrete ≥9
Time to first rescue analgesia | 24 hours post operative
  time to first demand for rescue analgesia
Bowel recovery (first flatus) | 48 hours post operative
  Time in hours from completion of surgery until the patient passes first flatus, representing bowel recovery.
Ambulation tolerance | 48 hours post operative
  Assessment of the patient's ability to ambulate, measured as distance walked in feet or meters within specified postoperative periods.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Aldrete, J. A. (1995). The post-anesthesia recovery score revisited. Journal of Clinical Anesthesia, *7*(1), 89-91. — https://doi.org/10.1016/0952-8180(94)00001-K
- See also: .National Institutes of Health. HEAL Initiative: Preventing Opioid Use Disorder After Surgery. NIH Guide NOT-DA-22-052. 2022. — https://grants.nih.gov/grants/guide/notice-files/NOT-DA-22-052.html
- See also: . Huskisson, E. C. (1974). Measurement of pain. The Lancet, *304*(7889), 1127-1131. — https://doi.org/10.1016/S0140-6736(74)90884-8